CLINICAL TRIAL: NCT05432700
Title: Randomised Clinical Trial for Evaluation of the Effectiveness of a Mobile Application in the Improvement of Breastfeeding up to 6 Months
Brief Title: Evaluation of the Effectiveness of LactApp
Acronym: COMLACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Francisco Javier Soriano-Vidal, Collaborating researcher., Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UGP-20-100
Record Dates: First submitted 2022-05-03; First posted 2022-06-27 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Breast Feeding
Keywords: Breast Feeding; Lactation; Mobile Applications; Software Validation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: After reading the patient information sheet and accepting the informed consent, they will be registered on the Breastfeeding Study web platform and included in one of the groups (intervention/control) through a randomisation process. Women will be selected during the third trimester of pregnancy at the surgery and during the midwifery routine care in each health department. Women in the intervention group will be provided with information on how to download the free LactApp® app for iOS and Android.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: usual clinical practice. (No Intervention): The women will receive an initial Health Literacy Survey (HLS-EU-Q16) via the email account registered on the platform. From this point until birth, no further notifications will be sent.
  Subsequently, reminders will be planned via email to obtain information on BF follow-up, avoiding providing any extra information on BF and, where appropriate, referring to the BF support services available in their area, following a standard clinical practice. During pregnancy, the pregnancy programme of the local and national government provides parenting education and breastfeeding workshops, with various manuals published.
  Surveys adapted to this group will be sent out at birth, at 15 days, 6 weeks, 3 and 6 months. The variables to be collected are socio-demographic, related to health literacy, obstetric-neonatal, and breastfeeding variables.
- Intervention group: LactApp (Experimental): From the initial registration in LactApp during the third trimester, women will be able to consult all the information available in the application. The women will receive an initial Health Literacy Survey (HLS-EU-Q16), from this point until birth, no further notifications will be sent. A reminder schedule will be made via email to obtain information on the follow-up of the BF.
  LactApp® works as a self-administered questionnaire based on decision trees constructed with questions and answers developed by professional breastfeeding experts, supported by scientific evidence and updated official health recommendations. In addition, the app will remind them of the topics according to the estimated date of birth provided. Surveys adapted to this group will be sent out at birth, at 15 days, 6 weeks, 3 and 6 months. The variables to be collected are socio-demographic, related to health literacy, obstetric-neonatal, and breastfeeding variables.
  Interventions: Other: LactApp

INTERVENTIONS:
Other: LactApp — LactApp® provides personalised answers that can be arrived at through different pathways, which vary according to the profile of the user and the options she selects, allowing data sampling through an Ecological Momentary Assessment.
  The app will remind of:
  The first month: baby's breastfeeding position, frequency of feeds, number and consistency of stools, general breast care, average weight gain; in mothers who gave some supplementation, advice and support for them to try re-breastfeeding.
  From the second to the third month: advice on expressing milk to create a reserve just in case they went back to work or had to be absent from home for a day, instructions on how to handle and preserve milk.
  From the fourth to the sixth month: indications to use the stored milk (if it was created) and techniques for administering it to the infant, the importance of maintaining the EBF and the inadvisability of offering other types of milk or food.
  Arms: Intervention group: LactApp

SUMMARY:
The study aims to determine the influence of an intervention in women based on a free mobile application (LactApp®) on maintaining breastfeeding (BF) up to 6 months postpartum. This is an experimental, multicentre, prospective study with a control group comparing the duration of BF. It will be carried out in the Health Departments of La Ribera, Xàtiva-Ontinyent, Castelló and Extremadura in 2021, 2022 and 2023. Women will be randomly assigned to each of the parallel groups. In the control group, the usual clinical practice will be followed from the third trimester of gestation to promote BF. In the intervention group, the woman, in addition to the usual clinical practice, will use a free mobile app: LactApp®, from the third trimester until 6 months postpartum. The type of breastfeeding at birth, 15 days, 3 and 6 months postpartum, and the causes of cessation of BF in both groups will be monitored. Socio-demographic data and the woman's reported outcomes will be collected during the pregnancy, birth, and postpartum process. The mobile app will report data on use, topics consulted and usage times. The null hypothesis is that the ¨LactApp®¨ mobile application does not improve breastfeeding maintenance at 6 months postpartum compared to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- Women who show a desire to breastfeed during the third trimester of pregnancy, with a command of Spanish, and whose birth will occur in one of the participating hospitals.

Exclusion Criteria:

* Not having a mobile device with an internet connection.
* Newborns of less than 37 weeks of gestation or with congenital malformations. malformations.
* Twin or multiple pregnancies, pregnancies admitted to neonatal care, or postpartum complications result in the mother being admitted to the intensive care unit.
* Women who do not respond respond to the automatic messages provided by the platform.
* In the intervention group, the non-installation of the mobile app Lactapp® mobile application.
* Women who have used the Lactapp® application on their own initiative will be excluded from the control group.

Ages: 16 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Use mobile app LactApp and Breastfeeding ratio. | 6 months since date of birth.
  Rate of breastfeeding at 6 months postpartum for women who have used the mobile app LactApp compared with women in routine care arm.

SECONDARY OUTCOMES:
Prevalence of BF. | 6 months since date of birth.
  Prevalence of breastfeeding at discharge and breastfeeding at 6 months postpartum.
Reported causes of BF cessation. | 6 months since date of birth.
  Women's reported causes of breastfeeding cessation, frequency of reported causes o breastfeeding cessation, and the length of breastfeeding up to six months postpartum.
Acceptability in the use of the LactApp mobile application. | 6 months since date of birth.
  Evaluation by the participants of the convenience, acceptability and user-friendliness of the mobile application. No personal information derived from the use of the mobile application will be collected.
HLS-EU-Q16 health literacy measurement and BF | 6 months since date of birth.
  HLS-EU-Q16 instrument will be used as a screening tool to evaluate the woman's health literacy level against the early cessation of BF. It assesses the health literacy level in the population through a series of 16 items measured on a Likert-type scale from "very easy" to "very difficult". It is a single-factor scale with an internal consistency of 0.982 in the Spanish population, measured by Cronbach's alpha and McDonald's omega.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Vila-Candel, PhD, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Hospital La Ribera, Alzira, Valencia, Spain

REFERENCES:
- [Derived] Mena-Tudela D, Soriano-Vidal FJ, Vila-Candel R, Quesada JA, Aguilar L, Franco-Antonio C. Effect of Mobile-Based Counselling on Breastfeeding in Spain: A Randomized Controlled Trial Protocol (COMLACT Study). Healthcare (Basel). 2023 May 15;11(10):1434. doi: 10.3390/healthcare11101434. PMID 37239720